CLINICAL TRIAL: NCT00952419
Title: Immunogenicity and Safety of Multiple Formulations of an A/H1N1 Pandemic Vaccine in Healthy Subjects Aged 6 Months to 9 Years
Brief Title: A Study of Different Formulations of an A/H1N1 Pandemic Vaccine in Healthy Children Aged 6 Months to 9 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FUF15; UTN: U1111-1111-4713
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2011-07-11 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Influenza; Swine-origin A/H1N1 Influenza
Keywords: Influenza; Pandemic Flu; Swine-origin A/H1N1 Influenza; Children
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A/H1N1 Vaccine Group 1 (Experimental): Participants will receive A/H1N1 vaccine formulation 1
  Interventions: Biological: Monovalent Subvirion A/H1N1 Influenza vaccine
- A/H1N1 Vaccine Group 2 (Experimental): Participants will receive A/H1N1 vaccine formulation 2
  Interventions: Biological: Monovalent Subvirion A/H1N1 Influenza vaccine
- Placebo Group (Placebo Comparator): Participants will receive a placebo vaccine
  Interventions: Biological: Normal saline solution (placebo)

INTERVENTIONS:
Biological: Monovalent Subvirion A/H1N1 Influenza vaccine — 0.5 mL, Intramuscular Day 0 and Day 21 (3 to 9 years); 0.25 mL, Intramuscular on Day 0 and Day 21 (6 months to 35 Months)
  Arms: A/H1N1 Vaccine Group 1
Biological: Monovalent Subvirion A/H1N1 Influenza vaccine — 0.5 mL, Intramuscular Day 0 and Day 21 (3 to 9 years); 0.25 mL, Intramuscular on day 0 and Day 21 (6 months to 35 Months)
  Arms: A/H1N1 Vaccine Group 2
Biological: Normal saline solution (placebo) — 0.5 mL, Intramuscular Day 0 and Day 21 (3 to 9 years); 0.25 mL, Intramuscular on day 0 and Day 21 (6 months to 35 Months)
  Arms: Placebo Group

SUMMARY:
The purpose of the study is to evaluate different doses of the Influenza A/H1N1 pandemic vaccine in toddlers and children.

Primary Objectives:

* To describe the immunogenicity of the candidate vaccines after each injection.
* To describe the safety of the candidate vaccines after each injection.

DETAILED DESCRIPTION:
Participants will receive two injections of their randomized vaccine on Day 0 and Day 21, respectively.

ELIGIBILITY:
Inclusion Criteria :

All subjects:

* Provision of Informed Consent Form signed by the subject's parent(s)/legal representative (and by an independent witness if required by local regulations). In addition, provision of Assent Form signed by subjects aged 7 to 9 years
* Subject and parent/guardian are able to attend all scheduled visits and to comply with all trial procedures

Subjects aged 3 to 9 years:

* Healthy children aged 3 to 9 years on the day of inclusion

Subjects aged 6 to 35 months:

* Healthy infants and toddlers aged 6 to 35 months on the day of inclusion
* Born at full term of pregnancy (≥ 37 weeks) and with a birth weight ≥ 2.5 kg

Exclusion Criteria :

* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination
* Planned receipt of any vaccine prior to the Day 42 blood sample
* Receipt of blood or blood-derived products in the past 3 months which might interfere with the assessment of immune response
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months, or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis B surface antigen, or Hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances
* Self reported thrombocytopenia contraindicating intramuscular (IM) vaccination
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion contraindicating IM vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Chronic illness that in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.
* Any confirmed case of influenza (including swine-origin A/H1N1 Influenza) since March 2009
* Personal or family history of Guillain-Barré syndrome
* Active neoplastic disease or a history of any hematologic malignancy
* Known seizure/epilepsy history and/or taking anti-seizure medication
* Receipt of psychiatric drugs. Subjects receiving a single antidepressant drug and stable for at least 3 months prior to enrollment, without decompensating symptoms will be allowed to enroll in the study
* Febrile illness (temperature ≥ 100.4°F [≥ 38.0°C]) or moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 474 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (19):
- United States (19):
  - Miami Beach, Florida
  - Marietta, Georgia
  - Woodstock, Georgia
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Maddisonville, Kentucky
  - Metairie, Louisiana
  - Las Vegas, Nevada
  - Rochester, New York
  - Hermitage, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Cranston, Rhode Island
  - Barnwell, South Carolina
  - Austin, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Orem, Utah
  - South Jordan, Utah
  - Springville, Utah

REFERENCES:
- [Result] Plennevaux E, Blatter M, Cornish MJ, Go K, Kirby D, Wali M, Reeves-Hoche MK, Denis M. Influenza A (H1N1) 2009 two-dose immunization of US children: an observer-blinded, randomized, placebo-controlled trial. Vaccine. 2011 Feb 11;29(8):1569-75. doi: 10.1016/j.vaccine.2010.12.116. Epub 2011 Jan 8. PMID 21219979
- [Derived] Plennevaux E, Sheldon E, Blatter M, Reeves-Hoche MK, Denis M. Immune response after a single vaccination against 2009 influenza A H1N1 in USA: a preliminary report of two randomised controlled phase 2 trials. Lancet. 2010 Jan 2;375(9708):41-8. doi: 10.1016/S0140-6736(09)62026-2. Epub 2009 Dec 15. PMID 20018365
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 06 August 2009 to 13 August 2009 at 19 US clinical centers.
Pre-assignment Details: A total of 474 participants who met the inclusion and exclusion criteria were enrolled, vaccinated, and included in data analysis.
Groups:
- A/H1N1 Vaccine Group 1: Participants who received a dose of 7.5 μg hemagglutinin intramuscularly on Day 1 and Day 21, respectively.
- A/H1N1 Vaccine Group 2: Participants who received a dose of 15 μg hemagglutinin intramuscularly on Day 1 and Day 21, respectively.
- Placebo Group: Participants who received a dose of placebo (saline) intramuscularly on Day 1 and Day 21, respectively.
Period: Overall Study
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Started | 215 | 208 | 51
Completed | 209 | 198 | 51
Not Completed | 6 | 10 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Protocol Violation | 3 | 7 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group | Total
Number analyzed (Participants) | 215 | 208 | 51 | 474
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 215 | 208 | 51 | 474
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 4.1 (2.8) | 4.3 (2.8) | 3.7 (2.7) | 4.2 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 99 | 24 | 234
  Male | 104 | 109 | 27 | 240
Region of Enrollment [Number; unit: participants]
  United States | 215 | 208 | 51 | 474

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Antibody Titers ≥ 10 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age 6 to 35 Months
Description: Pre- and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Pre- and post-vaccination antibody titers were assessed in the per-protocol population
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 92 | 87 | 23
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 10 1/dil | 5 | 2 | 0
  Post-Vaccination 1 (Day 21) Titers at ≥ 10 1/dil | 72 | 79 | 0
  Post-Vaccination 2 (Day 42) Titers at ≥ 10 1/dil | 90 | 87 | 1

2. Primary Outcome: Number of Participants With Antibody Titers ≥ 40 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age 6 to 35 Months
Description: Seroprotection: Antibody titer of ≥ 40 1/dil. Antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and Day 21 post-vaccination
Population: Antibody titers were assessed in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 92 | 87 | 23
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 40 1/dil | 5 | 2 | 0
  Post-Vaccination 1 (Day 21) Titers at ≥ 40 1/dil | 43 | 42 | 0
  Post-Vaccination 2 (Day 42) Titers at ≥ 40 1/dil | 84 | 86 | 1

3. Primary Outcome: Geometric Mean Titers (GMT) of Antibodies Against A/California (H1N1 Vaccine) Strain - Age 6 to 35 Months
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Antibody titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 92 | 87 | 23
Titers
  Pre-Vaccination 1 (Day 0) GMT | 5.99 [5.10 to 7.04] | 5.48 [4.84 to 6.20] | 5.00 [5.00 to 5.00]
  Post-Vaccination 1 (Day 21) GMT | 33.3 [23.8 to 46.5] | 45.1 [32.8 to 62.0] | 5.08 [4.92 to 5.24]
  Post-Vaccination 2 (Day 42) GMT | 368 [271 to 500] | 586 [451 to 763] | 5.64 [4.39 to 7.24]

4. Primary Outcome: Number of Participants With Antibody Titers ≥ 10 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age 3 to 9 Years
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and 21 days post-vaccination
Population: Pre- and post-vaccination antibody titers were assessed in the per-protocol population
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 98 | 91 | 24
Participants
  Pre-Vaccination 1(Day 0) Titers at ≥ 10 1/dil | 7 | 4 | 7
  Post-Vaccination 1 (Day 21) Titers at ≥ 10 1/dil | 91 | 88 | 8
  Post-Vaccination 2 (Day 42) Titers at ≥ 10 1/dil | 98 | 91 | 8

5. Primary Outcome: Number of Participants With Antibody Titers ≥ 40 1/Dilution (1/Dil) Against A/California (H1N1 Vaccine) Strain - Age 3 to 9 Years
Description: Seroprotection: Antibody titer ≥ 40 1/dil. Antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and Day 21 post-vaccination
Population: Pre- and post-vaccination antibody titers were assessed in the per-protocol population
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 98 | 91 | 24
Participants
  Pre-Vaccination 1 (Day 0) Titers at ≥ 40 1/dil | 5 | 3 | 5
  Post-Vaccination 1 (Day 21) Titers at ≥ 40 1/dil | 64 | 68 | 5
  Post-Vaccination 2 (Day 42) Titers at ≥ 40 1/dil | 95 | 90 | 6

6. Primary Outcome: Geometric Mean Titers (GMT) of Antibodies Against A/California (H1N1 Vaccine) Strain - Age 3 to 9 Years
Description: Pre-vaccination and post-vaccination antibody titers were determined by the hemagglutination inhibition (HAI) test.
Time Frame: Pre-vaccination (Day 0) and Day 21 post-vaccination
Population: Antibody titers were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 98 | 91 | 24
Titers
  Pre-Vaccination 1 (Day 0) GMT | 6.01 [5.20 to 6.94] | 5.54 [5.03 to 6.10] | 11.9 [6.17 to 22.9]
  Post-Vaccination 1 (Day 21) GMT | 74.8 [53.5 to 105] | 104 [77.1 to 140] | 12.1 [6.53 to 22.3]
  Post-Vaccination 2 (Day 42) GMT | 459 [348 to 605] | 586 [454 to 756] | 14.3 [7.02 to 29.3]

7. Primary Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction Following Vaccination - Age 6 to 23 Months
Description: Solicited Injection Site Reactions: Tenderness, erythema (redness), swelling, induration (hardening), ecchymosis (bruising). Solicited systemic reactions: Fever (temperature), vomiting, crying abnormal, drowsiness, appetite lost, irritability.
Time Frame: Days 0 to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants with available reaction data, intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 61 | 56 | 18
Participants
  Any Solicited Injection Site Reaction - Any Dose | 33 | 23 | 11
  Grade (Grd) 3 Injection Site Reaction - Any Dose | 1 | 1 | 0
  Any Tenderness - Post Dose 1 | 24 | 14 | 5
  Any Tenderness - Post Dose 2 | 19 | 11 | 7
  Any Tenderness - Any Dose | 28 | 20 | 10
  Grd 3 Tenderness-Crying or movement less, Any Dose | 0 | 1 | 0
  Any Erythema - Post Dose 1 | 13 | 4 | 1
  Any Erythema - Post Dose 2 | 12 | 5 | 2
  Any Erythema - Any Dose | 19 | 7 | 3
  Grade 3 Erythema (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Swelling - Post Dose 1 | 4 | 5 | 0
  Any Swelling - Post Dose 2 | 3 | 3 | 1
  Any Swelling - Any Dose | 6 | 6 | 1
  Grade 3 Swelling (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Induration - Post Dose 1 | 6 | 3 | 1
  Any Induration - Post Dose 2 | 4 | 3 | 0
  Any Induration - Any Dose | 6 | 5 | 1
  Grade 3 Induration (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Ecchymosis - Post Dose 1 | 3 | 3 | 0
  Any Ecchymosis - Post Dose 2 | 2 | 2 | 0
  Any Ecchymosis - Any Dose | 4 | 4 | 0
  Grade 3 Ecchymosis (≥ 5 cm) Any Dose | 1 | 0 | 0
  Any Solicited Systemic Reaction - Any Dose | 31 | 32 | 11
  Any Grade 3 Solicited Systemic Reaction - Any Dose | 3 | 4 | 0
  Any Fever - Post Dose 1 | 6 | 2 | 0
  Any Fever - Post Dose 2 | 0 | 5 | 1
  Any Fever - Any Dose | 6 | 6 | 1
  Grade 3 Fever ( ≥102.1 ºF or ≥39.0 ºC) - Any Dose | 0 | 1 | 0
  Any Vomiting - Post Dose 1 | 1 | 4 | 0
  Any Vomiting - Post Dose 2 | 2 | 3 | 0
  Any Vomiting - Any Dose | 3 | 6 | 0
  Grade 3 Vomiting (> 6 episodes/24 hr) Any Dose | 0 | 3 | 0
  Any Crying Abnormal - Post Dose 1 | 17 | 12 | 5
  Any Crying Abnormal - Post Dose 2 | 8 | 9 | 4
  Any Crying Abnormal - Any Dose | 20 | 14 | 7
  Grade 3 Crying Abnormal (>3 hr) Any Dose | 3 | 2 | 0
  Any Drowsiness - Post Dose 1 | 8 | 11 | 3
  Any Drowsiness - Post Dose 2 | 8 | 7 | 2
  Any Drowsiness - Any Dose | 11 | 11 | 3
  Grade 3 Drowsiness (Sleeps most of time) Any Dose | 0 | 1 | 0
  Any Appetite Lost - Post Dose 1 | 8 | 12 | 3
  Any Appetite Lost - Post Dose 2 | 5 | 9 | 3
  Any Appetite Lost - Any Dose | 10 | 14 | 4
  Grd 3 Appetite Lost (Refused 3 meals) Any Dose | 0 | 1 | 0
  Any Irritability - Post Dose 1 | 23 | 22 | 7
  Any Irritability - Post Dose 2 | 14 | 17 | 6
  Any Irritability - Any Dose | 26 | 25 | 9
  Grade 3 Irritability (Inconsolable) Any Dose | 0 | 2 | 0

8. Primary Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction Following Vaccination - Age 24 to 35 Months
Description: Solicited Injection Site Reactions: Pain, erythema (redness), swelling, induration (hardening), ecchymosis (bruising). Solicited systemic reactions: Fever (temperature), headache, malaise (feeling unwell), myalgia (muscle aches and pains), shivering.
Time Frame: Days 0 to 7 post-vaccination
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 44 | 42 | 8
Participants
  Any Solicited Injection Site Reaction - Any Dose | 19 | 20 | 5
  Grade (Grd) 3 Injection Site Reaction - Any Dose | 0 | 2 | 0
  Any Pain - Post Dose 1 | 12 | 12 | 3
  Any Pain - Post Dose 2 | 10 | 16 | 2
  Any Pain - Any Dose | 17 | 19 | 3
  Grade 3 Pain (Incapacitating) - Any Dose | 0 | 2 | 0
  Any Erythema - Post Dose 1 | 5 | 7 | 3
  Any Erythema - Post Dose 2 | 3 | 9 | 1
  Any Erythema - Any Dose | 6 | 12 | 3
  Grade 3 Erythema (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Swelling - Post Dose 1 | 1 | 3 | 0
  Any Swelling - Post Dose 2 | 0 | 3 | 0
  Any Swelling - Any Dose | 1 | 4 | 0
  Grade 3 Swelling (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Induration - Post Dose 1 | 2 | 4 | 1
  Any Induration - Post Dose 2 | 1 | 3 | 1
  Any Induration - Any Dose | 2 | 6 | 1
  Grade 3 Induration (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Ecchymosis - Post Dose 1 | 1 | 3 | 2
  Any Ecchymosis - Post Dose 2 | 2 | 3 | 0
  Any Ecchymosis - Any Dose | 3 | 6 | 2
  Grade 3 Ecchymosis (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Solicited Systemic Reaction - Any Dose | 14 | 13 | 3
  Any Grade 3 Solicited Systemic Reaction - Any Dose | 1 | 2 | 1
  Any Fever - Post Dose 1 | 1 | 1 | 1
  Any Fever - Post Dose 2 | 3 | 1 | 0
  Any Fever - Any Dose | 4 | 2 | 1
  Grade 3 Fever (≥ 102.1 ºF or ≥ 39.0 ºC) -Any Dose | 1 | 1 | 1
  Any Headache - Post Dose 1 | 1 | 1 | 1
  Any Headache - Post Dose 2 | 0 | 1 | 1
  Any Headache - Any Dose | 1 | 2 | 1
  Grd 3 Headache (Prevents daily activity) Any Dose | 0 | 0 | 0
  Any Malaise - Post Dose 1 | 7 | 6 | 3
  Any Malaise - Post Dose 2 | 5 | 6 | 2
  Any Malaise - Any Dose | 10 | 9 | 3
  Grd 3 Malaise (Prevents daily activity) Any Dose | 1 | 1 | 0
  Any Myalgia - Post Dose 1 | 4 | 3 | 2
  Any Myalgia - Post Dose 2 | 0 | 2 | 2
  Any Myalgia - Any Dose | 4 | 5 | 2
  Grd 3 Myalgia (Prevents Daily Activity) Any Dose | 0 | 0 | 0
  Any Shivering - Post Dose 1 | 1 | 1 | 0
  Any Shivering - Post Dose 2 | 0 | 0 | 0
  Any Shivering - Any Dose | 1 | 1 | 0
  Grade 3 Shivering (Prevents activity) - Any Dose | 0 | 0 | 0

9. Primary Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction Following Vaccination - Age 3 to 9 Years
Description: as for outcome 8
Time Frame: Days 0 to 7 post vaccination
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Number analyzed (Participants) | 114 | 106 | 25
Participants
  Any Solicited Injection Site Reaction - Any Dose | 70 | 59 | 16
  Grade 3 Injection Site Reaction - Any Dose | 3 | 3 | 0
  Any Pain - Post Dose 1 | 48 | 42 | 12
  Any Pain - Post Dose 2 | 34 | 31 | 8
  Any Pain - Any Dose | 63 | 54 | 16
  Grade 3 Pain (Incapacitating) - Any Dose | 2 | 0 | 0
  Any Erythema - Post Dose 1 | 14 | 14 | 2
  Any Erythema - Post Dose 2 | 10 | 5 | 2
  Any Erythema - Any Dose | 19 | 15 | 2
  Grade 3 Erythema (≥ 5 cm) Any Dose | 1 | 1 | 0
  Any Swelling - Post Dose 1 | 5 | 10 | 1
  Any Swelling - Post Dose 2 | 5 | 3 | 0
  Any Swelling - Any Dose | 8 | 11 | 1
  Grade 3 Swelling (≥ 5 cm) Any Dose | 1 | 3 | 0
  Any Induration - Post Dose 1 | 7 | 8 | 4
  Any Induration - Post Dose 2 | 7 | 2 | 0
  Any Induration - Any Dose | 11 | 8 | 4
  Grade 3 Induration (≥ 5 cm) Any Dose | 1 | 0 | 0
  Any Ecchymosis - Post Dose 1 | 9 | 9 | 1
  Any Ecchymosis - Post Dose 2 | 6 | 4 | 1
  Any Ecchymosis - Any Dose | 13 | 11 | 2
  Grade 3 Ecchymosis (≥ 5 cm) Any Dose | 0 | 0 | 0
  Any Solicited Systemic Reaction - Any Dose | 51 | 38 | 12
  Any Grade 3 Solicited Systemic Reaction - Any Dose | 5 | 7 | 2
  Any Fever - Post Dose 1 | 2 | 1 | 1
  Any Fever - Post Dose 2 | 4 | 5 | 1
  Any Fever - Any Dose | 6 | 6 | 2
  Grade 3 Fever (≥ 102.1 ºF or ≥ 39.0 ºC) - Any Dose | 1 | 3 | 1
  Any Headache - Post Dose 1 | 15 | 11 | 5
  Any Headache - Post Dose 2 | 13 | 10 | 3
  Any Headache - Any Dose | 23 | 19 | 7
  Gr 3 Headache (Prevents daily activity) Any Dose | 0 | 4 | 0
  Any Malaise - Post Dose 1 | 18 | 12 | 7
  Any Malaise - Post Dose 2 | 16 | 14 | 5
  Any Malaise - Any Dose | 29 | 24 | 10
  Gr 3 Malaise (Prevents daily activity) Any Dose | 3 | 6 | 1
  Any Myalgia - Post Dose 1 | 19 | 9 | 1
  Any Myalgia - Post Dose 2 | 14 | 11 | 3
  Any Myalgia - Any Dose | 32 | 18 | 3
  Gr 3 Malaise (Prevents daily activity) Any Dose | 2 | 0 | 0
  Any Shivering - Post Dose 1 | 1 | 3 | 1
  Any Shivering - Post Dose 2 | 0 | 5 | 1
  Any Shivering - Any Dose | 1 | 8 | 2
  Grade 3 Shivering (Prevents activity) - Any Dose | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination to up to 6 months post-vaccination.
Arm/Group | A/H1N1 Vaccine Group 1 | A/H1N1 Vaccine Group 2 | Placebo Group
Serious Adverse Events (participants affected / at risk) | 1/219 | 0/204 | 1/51
Other Adverse Events (participants affected / at risk) | 110/219 | 104/204 | 27/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A/H1N1 Vaccine Group 1 (N=219) | A/H1N1 Vaccine Group 2 (N=204) | Placebo Group (N=51)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | A/H1N1 Vaccine Group 1 (N=219) | A/H1N1 Vaccine Group 2 (N=204) | Placebo Group (N=51)
Pyrexia (General disorders) | 10 | 12 | 1
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 22 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 29 | 22 | 4
Injection site pain (General disorders) | 80/156 | 73/145 | 19/33
Injectiuon site tenderness (General disorders) | 28/61 | 20/55 | 10/18
Injection site erythema (General disorders) | 44/217 | 34/201 | 8
Injection site swelling (General disorders) | 15/217 | 21/201 | 2
Injection site induration (General disorders) | 19/217 | 19/201 | 6
Injection site ecchymosis (General disorders) | 20/217 | 21/201 | 4
Pyrexia (Fever) (General disorders) | 16/217 | 14/200 | 4
Headache (Nervous system disorders) | 24/156 | 21/145 | 8/33
Malaise (General disorders) | 39/156 | 33/145 | 13/33
Myalgia (Musculoskeletal and connective tissue disorders) | 36/156 | 23/145 | 5/33
Shivering (General disorders) | 2/156 | 9/145 | 2/33
Vomiting (Gastrointestinal disorders) | 3/61 | 6/55 | 0/18
Crying abnormal (Psychiatric disorders) | 20/61 | 14/55 | 7/18
Drowsiness (Nervous system disorders) | 11/61 | 11/55 | 3/18
Appetite lost (Metabolism and nutrition disorders) | 10/61 | 14/55 | 4/18
Irritability (Psychiatric disorders) | 26/61 | 25/55 | 9/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications